CLINICAL TRIAL: NCT03861208
Title: Assessing if Feelings of Hunger and Fullness Affect Learning in Children 3-4 Years Old
Brief Title: Hunger and Learning Study in Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Sibylle Kranz, PhD, RDN, Associate Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: SBS 2018007700
Record Dates: First submitted 2019-01-29; First posted 2019-03-04 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Hunger; Ingestive Behavior; Obesity; Food Preferences
MeSH Terms: conditions — Feeding Behavior; Obesity; Food Preferences | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diet (Experimental): high fiber high protein foods served in childcare centers are offered for meals and snacks
  Interventions: Other: diet
- usual diet (Other): foods representing the usual diet in childcare centers are offered for meals and snacks
  Interventions: Other: usual diet

INTERVENTIONS:
Other: diet — foods with high satiation (high protein and high fiber foods) are offered to modify children's hunger and fullness ratings postprandial
  Other Names: High protein high fiber
  Arms: diet
Other: usual diet — foods representing the usually provided foods at childcare are offered
  Arms: usual diet

SUMMARY:
This prospective random controlled cross-over intervention studies is designed to ascertain if children feel different levels of hunger and fullness before and after eating test meals consisting of high-satiety vs. usual foods and if the child's perceived hunger/fullness is related to their salivary ghrelin levels and a variety of learning outcomes. Data are collected at the Diet and Nutrition (DAN) laboratory on repeated study days (8am - 4 pm).

DETAILED DESCRIPTION:
The investigator's previous research has shown that preschoolers recognized changes in the feelings of hunger/fullness before and after a single test meal. If preschooler's feelings of hunger are associated with their ghrelin (hunger hormone) levels is not known. This study is designed to assess children's changes in feelings of hunger throughout the day (8 pm to 4 pm) and to measure both subjective feelings of hunger and salivary ghrelin levels before and after a standardized test meal (lunch).

An important secondary outcome related to children's feelings of hunger is their ability to learn. Currently, there is lack of data on the direct link between perceived hunger/fullness and learning processes. This study addresses these gaps using preschooler's perceived feelings of hunger and fullness (using a published 4-point scale (Kranz S.et al. "High-Protein and High-Dietary-Fiber Breakfasts Result in Equal Feelings of Fullness and Better Diet Quality in Low-Income Preschoolers Compared with Their Usual Breakfast" J Nutr doi: 10.3945/jn.116.234153, 2017) and a battery of learning tests (HTKS, KRISP, Stroop-style tasks, Woodcock Johnson vocabulary test, DCCS, and curisoty measures.)

ELIGIBILITY:
Inclusion Criteria:

* healthy children

Exclusion Criteria:

* no food allergies
* no medications that affect behavior/learning/appetite

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
hunger/fullness 120 minutes postprandial using "children's hunger scale" | change on hunger/fullness scale from pre-lunch to 2-hours post lunch
  hunger/fullness scale. change in children's perceived hunger and fullness on an age-appropriate scale: children respond to the question of "are you hungry or full" (coded hungry (1 or 2) or full (3 or 4)) followed by "are you very hungry( or full) or just a little hungry (or full)" coded as 1=very hungry, 2=a little hungry, 3- a little full, 4=very full, thus leading to a 4-point likert scale (from 1 to 4 with 1 being "very hungry" and 4 being "very full"). The development of the scale and its use are published by Kranz S. et al, Journal of Nutrition, 2017.
salivary ghrelin levels | change in salivary ghrelin from pre-lunch to 2-hours post lunch
  change in salivary ghrelin levels will be measured

SECONDARY OUTCOMES:
learning (working memory) | change from pre-lunch to 2-hours post lunch
  Head Toes Knee and Shoulders test
physical activity level | through study completion, on average of 8 weeks
  children will wear accelerators while at the laboratory ( 8 pm to 4 pm) to calculate average activity level across the 4 study days
liking of food | through study completion, on average of 8 weeks
  children will rate the foods provided using an age-appropriate visual (smiley faces) response coded as "like"(smiling face), "neutral" (face with straight line as mouth(, and "don't like" (face with tongue sticking out).
anthropometric data | at baseline
  measured height and weight to calculate CDC BMI-for-age percentiles of body weight status
systolic and diastolic blood pressure | through study completion, on average of 8 weeks
  measured systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Kranz, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Kranz S, Brauchla M, Campbell WW, Mattes RD, Schwichtenberg AJ. High-Protein and High-Dietary Fiber Breakfasts Result in Equal Feelings of Fullness and Better Diet Quality in Low-Income Preschoolers Compared with Their Usual Breakfast. J Nutr. 2017 Mar;147(3):445-452. doi: 10.3945/jn.116.234153. Epub 2017 Jan 11. PMID 28077732
- [Background] Kranz S, Marshall YW, Wight A, Bordi PL, Kris-Etherton PM. Liking and consumption of high-fiber snacks in preschool-age children. Food Quality and Preference 22: 486-489, 2011.